CLINICAL TRIAL: NCT04858516
Title: Neoadjuvant Treatment With Palbociclib and Exemestane Plus Trastuzumab and Pyrotinib in ER-positive, HER2-positive Breast Cancer (neoPEHP): an Exploratory, Open-label, Multi-center Phase 2 Study
Brief Title: Neoadjuvant Treatment With Palbociclib and Exemestane Plus Trastuzumab and Pyrotinib in Estrogen Receptor (ER)-Positive, HER2-positive Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20201101.2
Record Dates: First submitted 2021-04-18; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Neoadjuvant Treatment for HER2-positive, ER-positive Breast Cancer
MeSH Terms: interventions — palbociclib; exemestane; Trastuzumab; pyrotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant treatment with palbociclib and exemestane plus trastuzumab and pyrotinib (Experimental)
  Interventions: Drug: palbociclib and exemestane plus trastuzumab and pyrotinib

INTERVENTIONS:
Drug: palbociclib and exemestane plus trastuzumab and pyrotinib — Neoadjuvant treatment with palbociclib and exemestane plus trastuzumab and pyrotinib in ER-positive, HER2-positive breast cancer

SUMMARY:
neoPEHP is a multicohort, open-label, exploratory, phase 2 study. Patients were eligible if they had previously untreated, histologically confirmed, unilateral, invasive, HER2-positive, ER-positive breast cancer and were suitable for neoadjuvant therapy. Patients were treated every 3 weeks with intravenous trastuzumab (8 mg/kg loading dose followed by 6 mg/kg) and oral pyrotinib (400 mg po QD) for six cycles plus oral palbociclib (125 mg once a day for 21 days in a 4-week cycle) and oral exemestane (25 mg po QD) every 4 weeks for 24 weeks. The primary endpoints was pathological complete response.

ELIGIBILITY:
Inclusion Criteria:

* We judged patients eligible for the first study cohort if they had previously untreated, histologically confirmed, unilateral, invasive, HER2-positive (3+ on immunohistochemistry or neu-amplified) and ER-positive (>10% of cells in the tumour expressing ER) breast cancer. Other inclusion criteria were age 18 years or older, Eastern Cooperative Oncology Group (ECOG) performance status of 1 or less, and tumour classified between cT1c and cT4a-d.

Exclusion Criteria:

* metastatic disease, bilateral breast cancer, other malignant disease, inadequate bone marrow or renal function, impaired liver function, impaired cardiac function, uncontrolled hypertension, pregnancy, and refusal to use contraception.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2021-04-30 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
pathological complete response(ypT0/is,ypN0, pCR) | 24 weeks
  defined as the absence of invasive tumor cells in breast and axilla, ypT0/is ypN0